CLINICAL TRIAL: NCT00067080
Title: A Randomized, Open Label, Phase II Study on Safety and Efficacy of Long Term Treatment of ICL670 Relative to Deferoxamine in Sickle Cell Disease Patients With Transfusional Hemosiderosis
Brief Title: Safety of ICL670 vs. Deferoxamine in Sickle Cell Disease Patients With Iron Overload Due to Blood Transfusions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A0109
Record Dates: First submitted 2003-08-11; First posted 2003-08-13 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Anemia, Sickle Cell
Keywords: Sickle cell disease; iron overload; deferoxamine; hemosiderosis
MeSH Terms: conditions — Anemia, Sickle Cell; Iron Overload; Hemosiderosis | interventions — Deferasirox; Deferoxamine

ARMS (1):
- ICL670 + deferoxamine (Experimental)
  Interventions: Drug: ICL670, deferoxamine

INTERVENTIONS:
Drug: ICL670, deferoxamine
  Other Names: deferasirox

SUMMARY:
The purpose of this study is to determine if the new orally active iron chelator, ICL670, is as safe as deferoxamine in preventing accumulation of iron in the body while a patient is undergoing repeated blood transfusions.

DETAILED DESCRIPTION:
Patients who require repeated blood transfusions accumulate iron in the body as blood cells contain iron and there is no natural body mechanism to eliminate it. After a while the iron levels get high enough to be toxic to the body. The current therapy of choice is deferoxamine which does a good job of removing excess iron, but is difficult to administer. Deferoxamine requires subcutaneous (under the skin) infusions over 4 to 8 hours nightly 3 to 7 nights per week. In addition to the need to wear an infusion pump nightly, adverse reactions around the site of the injection are frequent.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 2 years
* Sickle cell disease patients already treated with or suitable for treatment with deferoxamine 20 to 40 mg/kg/day
* Serum ferritin greater than 1000 mg/ml
* Liver iron content greater than 2 mg iron/g dw assessed by means of superconducting quantum interference device (SQUID) for patients who receive simple transfusions and greater than 5 mg iron/ g dw for patients who receive exchange transfusions or who have a history of intermittent blood transfusion.
* Regular transfusion aimed at maintaining % Hb A above 50% or a previous history of simple transfusion being the recipient of at least 20 units of packed red blood cells.

Exclusion Criteria:

* Chronic anemias other than sickle cell disease
* Documented toxicity to deferoxamine
* Elevated liver enzymes in the year preceeding enrollment
* Active hepatitis B or hepatitis C
* HIV seropositivity
* Elevated serum creatinine or significant proteinuria
* History of nephrotic syndrome
* Uncontrolled systemic hypertension
* Fever and other signs/symptoms of infection within 10 days prior to the start of the study
* Presence of clinically relevant cataract or previous history of clinically relevant ocular toxicity related to iron chelation
* Second or third degree AV block, clinically relevant Q-T interval prolongation, or patients requiring digoxin or other drugs that prolong the Q-T interval (other than beta-adrenergic receptor blocking agents).
* Diseases (cardiovascular, renal, hepatic, etc.) that would prevent the patient from undergoing any of the treatment options
* Psychiatric or addictive disorders that would prevent the patient from giving informed consent
* History of drug or alcohol abuse within the 12 months prior to the study
* Pregnant or breast feeding patients
* Patients treated with systemic investigational drugs within 4 weeks or topical investigational drugs within 7 days before the start of the study
* Patients who require concomitant therapy with hydroxyurea
* Any surgical or medical condition that might significantly alter the absorption, distribution, metabolism or excretion of any drug, such as gastrointestinal disease or major surgery, renal disease, difficulty voiding or urinary obstruction, or impaired pancreatic function
* Non-compliant or unreliable patients
* Patients unable to undergo any study procedures such as the hearing or eye tests, or the liver echocardiography
* Patients unable to undergo SQUID examination

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2003-05; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of multiple doses of ICL670 | 1 year

SECONDARY OUTCOMES:
Estimate the absolute and relative change of liver iron content (LIC) and total body iron excretion (TBIE) | at baseline, after 24 weeks and at 1year (end of study)
Evaluate the pharmacokinetics | 24 hours post-dose @ 4, 12, 24 and 52 weeks
Evaluate the relationship between pharmacokinetics, pharmacodynamics and safety variables | at 24 and 52 weks pre-dose
Evaluate the relationship between hepatic iron and potential surrogate markers | at screen, at washout, then every 2 weeks for the first 12 weeks followed by every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (34):
- United States (34):
  - U. of S. Alabama Medical Center, Mobile, Alabama
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital & Research Center, Oakland, California
  - Colorado Sickle Cell Treatment and Research Center, Denver, Colorado
  - Howard University Hospital, Washington D.C., District of Columbia
  - Tampa Children's Hospital at St Joseph's, Tampa, Florida
  - Georgia Comprehensive Sickle cell Center, Grady Hospital, Atlanta, Georgia
  - Adult Sickle Cell Clinic, Medical College of Georgia, Augusta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Tulane University Sickle Cell Center, New Orleans, Louisiana
  - Children's Hospital, Department of Hematology/Oncology, New Orleans, Louisiana
  - Children's Hospital Boston, Division of Hematology/Oncology, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - NY Methodist Hospital, Brooklyn, New York
  - Weill Medical College of Cornell University, New York, New York
  - U. Of Rochester Medical Center, Rochester, New York
  - Sickle Cell Center, Montefiore Hospital, The Bronx, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Barrett Center, University of Cincinnati, Cincinnati, Ohio
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - James Cancer Hospital, Columbus, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Liberty Hematology Oncology Center, Columbia, South Carolina
  - Palmetto Health Clinical Trials, Columbia, South Carolina
  - Santee Hematology/Oncology, Sumter, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas
  - Scott and White Memorial Hospital & Clinics, Temple, Texas
  - Children's Hospital of the King's Daughter, Norfolk, Virginia

REFERENCES:
- [Result] Vichinsky E, Onyekwere O, Porter J, Swerdlow P, Eckman J, Lane P, Files B, Hassell K, Kelly P, Wilson F, Bernaudin F, Forni GL, Okpala I, Ressayre-Djaffer C, Alberti D, Holland J, Marks P, Fung E, Fischer R, Mueller BU, Coates T; Deferasirox in Sickle Cell Investigators. A randomised comparison of deferasirox versus deferoxamine for the treatment of transfusional iron overload in sickle cell disease. Br J Haematol. 2007 Feb;136(3):501-8. doi: 10.1111/j.1365-2141.2006.06455.x. PMID 17233848
- See also: Results for CICL670A0109 from the Novartis Clinical Trials website — https://www.ncbi.nlm.nih.gov/pubmed/17233848